CLINICAL TRIAL: NCT04223427
Title: Effects of Directional Subthalamic Deep Brain Stimulation on Gait and Balance in Parkinson's Disease Patients - MApping Gait and Balance Issues With Current Shaping
Brief Title: Effects of Directional Subthalamic Deep Brain Stimulation on Gait and Balance in Parkinson's Disease Patients
Acronym: MAGIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/0427/HP
Record Dates: First submitted 2019-12-10; First posted 2020-01-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The order of the five STN-DBS stimulation conditions will be randomized and assessments will be performed blinded from the stimulation condition. The effects of STN DBS on gait recordings will be assessed in 5 different conditions: with single ring DBS (1), and with current shaping for DBS of the gait 'hot spot' (2), of the dorsal STN (3) of the ventral STN (4) and of the DBS of narrow fiber tracts (5). The first condition will always be the single ring DBS.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single ring STN-DBS (Active Comparator): The order of the five STN-DBS stimulation conditions will be randomized and assessments will be performed blinded from the stimulation condition. The effects of STN DBS on gait recordings will be assessed in 5 different conditions: with single ring DBS (1), and with current shaping for DBS of the gait 'hot spot' (2), of the dorsal STN (3) of the ventral STN (4) and of the DBS of narrow fiber tracts (5). The first condition will always be the single ring DBS.
  Interventions: Procedure: Directional and single ring STN-DBS on gait
- Directional STN-DBS (Experimental): The order of the five STN-DBS stimulation conditions will be randomized and assessments will be performed blinded from the stimulation condition. The effects of STN DBS on gait recordings will be assessed in 5 different conditions: with single ring DBS (1), and with current shaping for DBS of the gait 'hot spot' (2), of the dorsal STN (3) of the ventral STN (4) and of the DBS of narrow fiber tracts (5). The first condition will always be the single ring DBS.
  Interventions: Procedure: Directional and single ring STN-DBS on gait

INTERVENTIONS:
Procedure: Directional and single ring STN-DBS on gait — Surgery for STN-DBS and STN-LFP recordings during gait initiation (M1): 15 days
  * Surgery for STN-DBS electrodes implantation
    * Placement of stimulation electrodes according to the usual procedure, including a MRI with contrast product
    * Intraoperative electrophysiological recordings
    * Intraoperative clinical evaluation
    * Intraoperative identification of the electrodes and final position with X-Ray
    * Post-operative 3D helical TDM without iode injection
  * STN-LFP recordings during gait initiation performed 3 to 5 days after surgery
  * Placement of the neurostimulator (5 days after surgery)
  * Acute testing of STN-DBS for first parameters setting programming
  Follow-up of the patient with outpatient visits as usually performed in PD patients operated for STN-DBS with progressive adaptation of parameters settings using single-ring stimulation.
  Directional and single ring STN-DBS on gait (M7)

SUMMARY:
Deep brain stimulation of the NST is effective for cardinal motor signs in patients with idiopathic Parkinson's disease (IPD), its effects on gait disturbances, especially freezing of gait-FOG, and falls are variable from one patient to another, in part depending on the location of the NST-stimulating contact. The ability to change the shape of the current field, and thus the volume of activated tissue, with a directional stimulation electrode is a new treatment option for NSC SCP patients with Parkinson's disease. In this pilot research program, the main objective is to determine the impact of directional DBS on gait and balance issues for PD patients implanted in the STN, using previously described anatomical and functional data for gait disturbances to guide directional programming. Ten patients with Patients with severe form of Parkinson's disease eligible to deep brain stimulation of the subthalamic nucleus, will be included in two French sites.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years
2. Diagnosis of Parkinson's Disease; as defined by the United Kingdom Parkinson's Disease Society Brain Bank (UKPDSBB) criteria
3. Patients eligible for subthalamic bilateral deep brain stimulation (STN-DBS) according to local inclusion criteria;
4. Freezing of gait in the OFF-dopa condition with item 2.13 of the MDS-UPDRS > 0 in usual life;
5. Patient having read and understood the information letter and signed the Informed Consent Form
6. Patient affiliated with, or beneficiary of a social security category
7. Stability of others medical disorders or that do not interfere with the research protocol.
8. Woman of childbearing potential with effective contraception according to WHO definition (estrogen-progestin or intra-uterine device or tubal ligation) since at least 3 months (negative urinary pregnancy test at inclusion)

Exclusion Criteria:

1. Actual and severe psychiatric pathology or other neurological disorder
2. Dementia (MMS <24/30)
3. Contraindication to research MRI (without contrast product) such as claustrophobia, metallic splinters in the eyes, ferromagnetic foreign bodies close to nerve structures, cardiac, ORL and neurological devices not MRI compatible, wearing of osteosynthseis equipment prior to 1980, metal prostheses, bypass valves ventriculoperitoneal neurosurgery, tattoos containing iron particles…
4. Contraindication to surgery: hemostasis trouble, anticoagulants or antiagregants treatment, ongoing infection
5. Hypersensitivity to contrasts agents
6. Persons under guardianship, tutorship or any other administrative or judicial measure of deprivation of rights and liberty
7. Subject at the time of exclusion from other biomedical research or participating in any other biomedical research or therapeutic trial
8. Pregnant or parturient or lactating woman or lack of proven and effective contraception according to WHO definition (estrogen-progestin or intra-uterine device or tubal ligation) (for women of childbearing age)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Changes in the principal components analysis (PCA) of the gait initiation kinetics during gait initiation with cognitive interference | 7 months
  The primary endpoint will be the changes in Euclidian distance in the principal components analysis (PCA) of the gait initiation kinetics during gait initiation with cognitive interference (Go, No Go paradigm), reproducing at least partly situations where FOG occurred, between stimulation conditions (Varriale, Collomb-Clerc, et al., 2018).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de ROUEN, Rouen, France, France